CLINICAL TRIAL: NCT00295646
Title: Tamoxifen Versus Anastrozole, Alone or in Combination With Zoledronic Acid, in Premenopausal, Hormone Receptor-positive Breast Cancer Patients (Stage I, II)
Brief Title: Tamoxifen Versus Anastrozole, Alone or in Combination With Zoledronic Acid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: AstraZeneca (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG-12; CZOL 446 1B 01 (Other: Novartis); Zol-A-01 (Other: Novartis)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: Austrian Breast & Colorectal Cancer Study Group (ABCSG); 12; Phase 3; breast cancer; anastrozole; tamoxifen; zoledronic acid; premenopausal; hormone receptor-positive; Stage I; Stage II; bone mineral density; BMD; bisphosphonate; zoledronate
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Anastrozole; Zoledronic Acid; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AZ (Arimidex+Zoledronate) (Active Comparator): Study Drugs Arimidex (Anastrozole), Zometa (Zoledronate; zoledronic acid)
  Interventions: Drug: anastrozole; Drug: zoledronic acid; Other: goserelin
- TZ (Tamoxifen+Zoledronate) (Active Comparator): Study Drugs Nolvadex (Tamoxifen), Zometa (Zoledronate; zoledronic acid)
  Interventions: Drug: tamoxifen; Drug: zoledronic acid; Other: goserelin
- AC (Arimidex Control) (Active Comparator): Study Drug Arimidex (Anastrozole)
  Interventions: Drug: anastrozole; Other: goserelin
- TC (Tamoxifen Control) (Active Comparator): Study Drug Nolvadex (Tamoxifen)
  Interventions: Drug: tamoxifen; Other: goserelin

INTERVENTIONS:
Drug: tamoxifen — 20 mg/d
  Other Names: Nolvadex
  Arms: TC (Tamoxifen Control); TZ (Tamoxifen+Zoledronate)
Drug: anastrozole — 1 mg/d
  Other Names: Arimidex
  Arms: AC (Arimidex Control); AZ (Arimidex+Zoledronate)
Drug: zoledronic acid — 4 mg q6m
  Other Names: Zoledronate, Zometa
  Arms: AZ (Arimidex+Zoledronate); TZ (Tamoxifen+Zoledronate)
Other: goserelin — 3.6 mg goserelin subcutaneously every 28 days

SUMMARY:
The primary objective is, first, the comparison of tamoxifen and anastrozole and, second, the comparison of zoledronate added to standard adjuvant therapy with controls according to disease-free survival (DFS) in premenopausal patients with non-metastatic breast cancer treated with tamoxifen or anastrozole. To assess whether zoledronate added to standard adjuvant therapy can decrease or even prevent bone loss in patients treated with hormonal blockade combined with an antiestrogen or aromatase inhibitor.

DETAILED DESCRIPTION:
The trial is conducted as an open multi-center phase III study, in a two-factorial study design and according to Good Clinical Practice (GCP) guidelines. Patients will be randomly assigned to a total of 4 study groups in a 1:1:1:1 assignment ratio. Several stratification criteria will be used in order to ensure balanced distribution of known risk factors.

A total of 1.803 patients will be enrolled in 4 arms. Patients will either be treated with anastrozole (1mg daily for 3 years) or tamoxifen (20mg daily for 3 years), and will additionally receive either zoledronate (8mg q4 weeks for 3 years) or no zoledronate (arm A: Nolvadex alone; arm B: Nolvadex plus zoledronate; arm C: Arimidex alone; arm D: Arimidex plus zoledronate).

Zoledronate will be administered by i.v. injection at a dose of 4 mg/month for the treatment period of 3 years. Five Bone Mineral Density (BMD) measurements will be performed in a subgroup of patients (404 patients, enrolled in 3 centres).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal, hormone receptor-positive patient
* Histologically verified (minimally) invasive breast cancer, local radical treatment
* 0-9 involved axillary lymph nodes (≥ 10 histologically examined nodes)
* Tumor stage: pT1b-3, yT0 or yT1a

Exclusion Criteria:

* T1a, T4d, yT4; M1
* Previous breast tumor irradiation
* Previous or concurrent chemotherapy (except for preoperative chemotherapy)
* Serum creatinine > 1.5 x UNL or creatinine clearance < 60 ml/min

Ages: 19 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1803 (Actual)
Dates: Start 1999-06; Primary Completion 2008-03-27 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (72):
- Austria (62):
  - Hospital of Guessing, Güssing, Burgenland
  - Hospital Oberpullendorf, Oberpullendorf, Burgenland
  - Hospital Oberwart, Oberwart, Burgenland
  - State Hospital Klagenfurt, Surgery, Klagenfurt, Carinthia
  - State Hospital Klagenfurt, Klagenfurt, Carinthia
  - Hospital BHB St. Veit, Saint Veit A. D. Glan, Carinthia
  - Ordination Dr. Wette, Saint Veit A. D. Glan, Carinthia
  - State Hospital Villach, Villach, Carinthia
  - Privat Hospital Villach, Villach, Carinthia
  - State Hospital Wolfsberg, Wolfsberg, Carinthia
  - Hospital Hainburg, Hainburg an der Donau, Lower Austria
  - Hospital Klosterneuburg, Internal Medicine, Klosterneuburg, Lower Austria
  - Hospital Krems, Krems, Lower Austria
  - Hospital Melk, Melk, Lower Austria
  - Hospital Mistelbach, Mistelbach, Lower Austria
  - Hospital Mödling, Mödling, Lower Austria
  - Hospital Neunkirchen, Neunkirchen, Lower Austria
  - Hospital St. Poelten, Sankt Pölten, Lower Austria
  - Hospital Scheibbs, Scheibbs, Lower Austria
  - Hospital Tulln, Tulln, Lower Austria
  - Hospital Waidhofen/Thaya, Waidhofen an der Thaya, Lower Austria
  - Hospital of Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Kardinal Schwarzenberg'sches Hospital, Schwarzach, Salzburg
  - State Hospital Feldbach, Feldbach, Styria
  - Gynaegological Medical University of Graz, Graz, Styria
  - Medical University of Graz, Oncology, Graz, Styria
  - State Hospital Leoben, Leoben, Styria
  - State Hospital Rottenmann, Rottenmann, Styria
  - Brustgesundheitszentrum-Süd Institut / Dr. Thiel, Weiz, Styria
  - District Hospital Hall in Tirol, Hall in Tirol, Tyrol
  - Gynaegological Medical University Innsbruck, Innsbruck, Tyrol
  - District Hospital Kufstein, Kufstein, Tyrol
  - District Hospital Lienz, Lienz, Tyrol
  - Hospital St. Vinzenz, Zams, Tyrol
  - State Hospital Bad Ischl, Bad Ischl, Upper Austria
  - State Hospital Freistadt, Freistadt, Upper Austria
  - State Hospital Gmunden, Gmunden, Upper Austria
  - State Hospital Kirchdorf, Kirchdorf, Upper Austria
  - Hospital BHS Linz, Linz, Upper Austria
  - Hospital Elisabethinen Linz, Linz, Upper Austria
  - General Hospital Linz, Linz, Upper Austria
  - Hospital BHB Linz, Linz, Upper Austria
  - Ordination Dr. Pöstlberger, Linz, Upper Austria
  - Hospital BHS Ried, Ried, Upper Austria
  - State Hospital Rohrbach, Rohrbach, Upper Austria
  - State Hospital Schärding, Schärding, Upper Austria
  - State Hospital Steyr, Steyr, Upper Austria
  - State Hospital Voecklabruck, Internal Medicine, Vöcklabruck, Upper Austria
  - State Hospital Voecklabruck, Surgery Dept., Vöcklabruck, Upper Austria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - State Hospital Bregenz, Bregenz, Vorarlberg
  - State Hospital of Dornbirn, Dornbirn, Vorarlberg
  - State Hospital Feldkirch, Feldkirch, Vorarlberg
  - Paracelsus Medical University Salzburg - Oncology, Salzburg
  - Hospital BHB Vienna, Surgery, Vienna
  - Hospital Sanatorium Hera, Vienna
  - Medical University of Vienna, General Hospital, Gynaecology and Obstetrics, Vienna
  - Medical University of Vienna, General Hospital, Vienna
  - Medical University Vienna, General Hospital, Vienna
  - State Hospital Vienna-Hietzing, Vienna
  - Hanusch Hospital, Vienna
  - Wilheminenspital, Internal Medicin I, Vienna
- Germany (10):
  - Practice Dr. Marschner, Freiburg im Breisgau, Baden-Wurttemberg
  - Medical Care Center, Ulm, Baden-Wurttemberg
  - Klinikum St. Marien, Amberg, Bavaria
  - Med. University of Munich, Munich, Bavaria
  - Frauenklinik vom Roten Kreuz, Munich, Bavaria
  - Elisabeth-Hospital, Kassel, Hesse
  - Internal-haematological Practice Oldenburg, Oldenburg, Lower Saxony
  - General Hospital Gifhorn, Gifhorn, Saxony
  - Medical University Kiel, Kiel, Schleswig-Holstein
  - Vivantes-Klinikum Friedrichshain, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gnant M, Mlineritsch B, Luschin-Ebengreuth G, Kainberger F, Kassmann H, Piswanger-Solkner JC, Seifert M, Ploner F, Menzel C, Dubsky P, Fitzal F, Bjelic-Radisic V, Steger G, Greil R, Marth C, Kubista E, Samonigg H, Wohlmuth P, Mittlbock M, Jakesz R; Austrian Breast and Colorectal Cancer Study Group (ABCSG). Adjuvant endocrine therapy plus zoledronic acid in premenopausal women with early-stage breast cancer: 5-year follow-up of the ABCSG-12 bone-mineral density substudy. Lancet Oncol. 2008 Sep;9(9):840-9. doi: 10.1016/S1470-2045(08)70204-3. Epub 2008 Aug 19. PMID 18718815
- [Background] Gnant MF, Mlineritsch B, Luschin-Ebengreuth G, Grampp S, Kaessmann H, Schmid M, Menzel C, Piswanger-Soelkner JC, Galid A, Mittlboeck M, Hausmaninger H, Jakesz R; Austrian Breast and Colorectal Cancer Study Group. Zoledronic acid prevents cancer treatment-induced bone loss in premenopausal women receiving adjuvant endocrine therapy for hormone-responsive breast cancer: a report from the Austrian Breast and Colorectal Cancer Study Group. J Clin Oncol. 2007 Mar 1;25(7):820-8. doi: 10.1200/JCO.2005.02.7102. Epub 2006 Dec 11. PMID 17159195
- [Background] Gnant M, Mlineritsch B, Schippinger W, Luschin-Ebengreuth G, Postlberger S, Menzel C, Jakesz R, Seifert M, Hubalek M, Bjelic-Radisic V, Samonigg H, Tausch C, Eidtmann H, Steger G, Kwasny W, Dubsky P, Fridrik M, Fitzal F, Stierer M, Rucklinger E, Greil R; ABCSG-12 Trial Investigators; Marth C. Endocrine therapy plus zoledronic acid in premenopausal breast cancer. N Engl J Med. 2009 Feb 12;360(7):679-91. doi: 10.1056/NEJMoa0806285. PMID 19213681
- [Background] Gnant M, Dubsky P, Fitzal F, Blaha P, Schoppmann S, Steger G, Marth C, Samonigg H, Huttner K, Fohler H, Ruecklinger E, Jakesz R, Greil R; Austrian Breast and Colorectal Cancer Study Group. Maintaining bone density in patients undergoing treatment for breast cancer: is there an adjuvant benefit? Clin Breast Cancer. 2009 Jun;9 Suppl 1:S18-27. doi: 10.3816/CBC.2009.s.002. PMID 19561003
- [Background] Gnant M. Can oral bisphosphonates really reduce the risk of breast cancer in healthy women? J Clin Oncol. 2010 Aug 1;28(22):3548-51. doi: 10.1200/JCO.2010.29.6327. Epub 2010 Jun 21. No abstract available. PMID 20567005
- [Background] Gnant M, Mlineritsch B, Stoeger H, Luschin-Ebengreuth G, Heck D, Menzel C, Jakesz R, Seifert M, Hubalek M, Pristauz G, Bauernhofer T, Eidtmann H, Eiermann W, Steger G, Kwasny W, Dubsky P, Hochreiner G, Forsthuber EP, Fesl C, Greil R; Austrian Breast and Colorectal Cancer Study Group, Vienna, Austria. Adjuvant endocrine therapy plus zoledronic acid in premenopausal women with early-stage breast cancer: 62-month follow-up from the ABCSG-12 randomised trial. Lancet Oncol. 2011 Jul;12(7):631-41. doi: 10.1016/S1470-2045(11)70122-X. Epub 2011 Jun 5. PMID 21641868
- [Background] Gnant M. Zoledronic acid in breast cancer: latest findings and interpretations. Ther Adv Med Oncol. 2011 Nov;3(6):293-301. doi: 10.1177/1758834011420599. PMID 22084643
- [Background] Pfeiler G, Konigsberg R, Fesl C, Mlineritsch B, Stoeger H, Singer CF, Postlberger S, Steger GG, Seifert M, Dubsky P, Taucher S, Samonigg H, Bjelic-Radisic V, Greil R, Marth C, Gnant M. Impact of body mass index on the efficacy of endocrine therapy in premenopausal patients with breast cancer: an analysis of the prospective ABCSG-12 trial. J Clin Oncol. 2011 Jul 1;29(19):2653-9. doi: 10.1200/JCO.2010.33.2585. Epub 2011 May 9. PMID 21555684
- [Background] Ressler S, Mlineritsch B, Greil R. Zoledronic acid for adjuvant use in patients with breast cancer. Expert Rev Anticancer Ther. 2011 Mar;11(3):333-49. doi: 10.1586/era.11.13. PMID 21417849
- [Background] Hadji P, Coleman R, Gnant M, Green J. The impact of menopause on bone, zoledronic acid, and implications for breast cancer growth and metastasis. Ann Oncol. 2012 Nov;23(11):2782-2790. doi: 10.1093/annonc/mds169. Epub 2012 Jun 22. PMID 22730099
- [Background] Rugani P, Luschin G, Jakse N, Kirnbauer B, Lang U, Acham S. Prevalence of bisphosphonate-associated osteonecrosis of the jaw after intravenous zoledronate infusions in patients with early breast cancer. Clin Oral Investig. 2014;18(2):401-7. doi: 10.1007/s00784-013-1012-5. Epub 2013 Jun 10. PMID 23749244
- [Background] Gnant M, Mlineritsch B, Stoeger H, Luschin-Ebengreuth G, Knauer M, Moik M, Jakesz R, Seifert M, Taucher S, Bjelic-Radisic V, Balic M, Eidtmann H, Eiermann W, Steger G, Kwasny W, Dubsky P, Selim U, Fitzal F, Hochreiner G, Wette V, Sevelda P, Ploner F, Bartsch R, Fesl C, Greil R; Austrian Breast and Colorectal Cancer Study Group, Vienna, Austria. Zoledronic acid combined with adjuvant endocrine therapy of tamoxifen versus anastrozol plus ovarian function suppression in premenopausal early breast cancer: final analysis of the Austrian Breast and Colorectal Cancer Study Group Trial 12. Ann Oncol. 2015 Feb;26(2):313-20. doi: 10.1093/annonc/mdu544. Epub 2014 Nov 17. PMID 25403582
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Adjuvant bisphosphonate treatment in early breast cancer: meta-analyses of individual patient data from randomised trials. Lancet. 2015 Oct 3;386(10001):1353-1361. doi: 10.1016/S0140-6736(15)60908-4. Epub 2015 Jul 23. PMID 26211824
- [Background] Lipton A, Gnant M, Aapro M. Managing aromatase inhibitor-associated bone loss in breast cancer. Womens Health (Lond). 2007 Jul;3(4):441-8. doi: 10.2217/17455057.3.4.441. PMID 19804020
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Beltran-Bless AA, Clemons MJ, Fesl C, Greil R, Pond GR, Balic M, Vandermeer L, Bjelic-Radisic V, Singer CF, Steger GG, Helfgott R, Egle D, Solkner L, Gampenrieder SP, Kacerovsky-Strobl S, Suppan C, Ritter M, Rinnerthaler G, Pfeiler G, Fohler H, Hlauschek D, Hilton J, Gnant M. Does the number of 6-monthly adjuvant zoledronate infusions received affect treatment efficacy for early breast cancer? A sub-study of ABCSG-12. Eur J Cancer. 2023 Feb;180:108-116. doi: 10.1016/j.ejca.2022.12.003. Epub 2022 Dec 10. PMID 36592505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was randomized June 17, 1999, the last patient was randomized May 17, 2006. Randomization took place in 66 Austrian and 10 German clinical sites. In total, 1.803 patients were enrolled.
Period: Overall Study
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
Started | 450 | 450 | 453 | 450
Completed | 415 | 409 | 403 | 405
Not Completed | 35 | 41 | 50 | 45
Not completed — Protocol Violation | 18 | 20 | 20 | 18
Not completed — Withdrawal by Subject | 8 | 9 | 11 | 14
Not completed — Lost to Follow-up | 0 | 5 | 1 | 5
Not completed — Death | 9 | 7 | 18 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control) | Total
Number analyzed (Participants) | 450 | 450 | 453 | 450 | 1803
Age, Continuous [Median (Full Range); unit: years] | 44 [28 to 56] | 45 [27 to 54] | 44 [25 to 58] | 45 [27 to 56] | 45 [25 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 450 | 450 | 453 | 450 | 1803
  Male | 0 | 0 | 0 | 0 | 0
pT-stage [Count of Participants; unit: Participants] — The pathologic T-stage (pT) describes the categories of tumor size: pT1: <2 cm, pT2: 2 to 5 cm, pT3: > 5 cm.
  Participants
    pT1 | 343 | 339 | 352 | 341 | 1375
    pT2/pT3 | 98 | 97 | 93 | 98 | 386
    Unknown | 9 | 14 | 8 | 11 | 42
pN-stage [Count of Participants; unit: Participants] — The pathologic N-stage (pN) describes the categories of affected lymph nodes: negative: no lymph node affected, positive: at least one lymph node affected.
  Participants
    Negative | 304 | 298 | 304 | 305 | 1211
    Positive | 137 | 138 | 141 | 134 | 550
    Unknown | 9 | 14 | 8 | 11 | 42
Histologic grade [Count of Participants; unit: Participants] — The histologic grade describes to which extent the cancer cells and their arrangement look look like normal cells. Grade 1 (G1): well-differentiated, cells look more like normal breast tissue; Grade (G2): moderately differentiated; Grade (G3): poorly differentiated; GX: grade cannot be assessed.
  Participants
    G1/G2 | 341 | 347 | 347 | 346 | 1381
    G3 | 93 | 85 | 89 | 85 | 352
    GX | 7 | 4 | 9 | 8 | 28
    Unknown | 9 | 14 | 8 | 11 | 42
Estrogen receptor status [Count of Participants; unit: Participants]
  Negative | 17 | 20 | 14 | 16 | 67
  Positive | 424 | 416 | 431 | 423 | 1694
  Unknown | 9 | 14 | 8 | 11 | 42
Progesterone receptor status [Count of Participants; unit: Participants]
  Negative | 36 | 32 | 35 | 40 | 143
  Positive | 405 | 404 | 409 | 399 | 1617
  Unknown | 9 | 14 | 9 | 11 | 43
Preoperative chemotherapy [Count of Participants; unit: Participants]
  No | 386 | 382 | 389 | 379 | 1536
  Yes | 26 | 23 | 23 | 25 | 97
  Unknown | 38 | 45 | 41 | 46 | 170

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Anastrozole vs Tamoxifen in Premenopausal Patients With Non-metastatic Breast Cancer With Respect to Disease-free Survival (DFS)
Description: DFS is defined as time from randomization to first occurrence of a local, regional, or distant recurrence, second primary carcinoma (including contralateral breast cancer), or death from any cause
Time Frame: Time from randomization to the analysis data cut-off date when 124 DFS events had occurred. On the analysis data cut-off date, maximum time on study per patient was 102 months.
Population: Intent-to-treat population: All participants assigned to one of the four treatment arms were included in the analysis
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
Number analyzed (Participants) | 450 | 450 | 453 | 450
years | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: AZ (Arimidex+Zoledronate) vs TZ (Tamoxifen+Zoledronate) vs AC (Arimidex Control) vs TC (Tamoxifen Control); To determine the effect of arimidex (AZ and AC) compared to tamoxifen (TZ and TC) in terms of disease-free survival. Disease-free survival (DFS) is defined as the time from randomization to the first occurrence of a local or regional recurrence, cancer in the contralateral breast, distant metastasis, second primary carcinoma, or death from any cause; Test type: Superiority — A two-sided significance level of 2.5% was used in this 2x2 factorial design of two primary endpoints according to the Bonferroni-Holm adjustment to control multiplicity; p = 0.59, Log Rank — Two-sided significance level of 2.5%, with the application of the Bonferroni-Holm adjustment for multiple comparisons; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.78 to 1.53] — From the Cox Proportional hazard model with endocrine treatment fitted as a covariate. A hazard ratio > 1.0 indicates a higher average event rate and a shorter disease-free time for arimidex relative to tamoxifen

2. Primary Outcome: Comparison of Zoledronate vs no Zoledronate in Premenopausal Patients With Non-metastatic Breast Cancer With Respect to Disease-free Survival (DFS)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Intent-to-treat population: All participants assigned to one of the four treatment arms were included in the analysis
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
Number analyzed (Participants) | 450 | 450 | 453 | 450
years | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: AZ (Arimidex+Zoledronate) vs TZ (Tamoxifen+Zoledronate) vs AC (Arimidex Control) vs TC (Tamoxifen Control); To determine the effect of Zoledronic Acid (AZ and TZ) compared to no Zoledronic Acid (AC and TC) in terms of disease-free survival. Disease-free survival (DFS) is defined as the time from randomization to the first occurrence of a local or regional recurrence, cancer in the contralateral breast, distant metastasis, second primary carcinoma, or death from any cause; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.01, Log Rank — Two-sided significance level of 2.5%, with the application of the Bonferroni-Holm adjustment for multiple comparisons; Cox Proportional Hazard = 0.64, 95% CI 2-sided [0.46 to 0.91] — From the Cox Proportional hazard model with Zoledronic Acid treatment fitted as a covariate. A hazard ratio < 1.0 indicates a lower average event rate and a longer disease-free time for Zoledronic Acid relative to no Zoledronic Acid

3. Secondary Outcome: Comparison of Anastrozole vs Tamoxifen in Premenopausal Patients With Non-metastatic Breast Cancer With Respect to Recurrence-free Survival (RFS)
Description: RFS is defined as time from randomization to first occurrence of a local, regional, or distant recurrence, second primary carcinoma (including contralateral breast cancer), or death from breast cancer
Time Frame: as for outcome 1
Population: Intent-to-treat population: All participants assigned to one of the four treatment arms were included in the analysis
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
Number analyzed (Participants) | 450 | 450 | 453 | 450
years | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: AZ (Arimidex+Zoledronate) vs TZ (Tamoxifen+Zoledronate) vs AC (Arimidex Control) vs TC (Tamoxifen Control); To determine the effect of arimidex (AZ and AC) compared to tamoxifen (TZ and TC) in terms of recurrence-free survival. Recurrence-free survival is defined as the time from randomization to the first occurrence of a local or regional recurrence, cancer in the contralateral breast, distant metastasis, second primary carcinoma, or death related to breast cancer; Test type: Superiority — No multiplicity adjustment was applied; p = 0.53, Log Rank; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.80 to 1.56] — From the Cox Proportional hazard model with endocrine treatment fitted as a covariate. A hazard ratio > 1.0 indicates a higher average event rate and a shorter recurrence-free time for arimidex relative to tamoxifen

4. Secondary Outcome: Comparison of Zoledronate vs no Zoledronate in Premenopausal Patients With Non-metastatic Breast Cancer With Respect to Recurrence-free Survival (RFS)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Intent-to-treat population: All participants assigned to one of the four treatment arms were included in the analysis
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
Number analyzed (Participants) | 450 | 450 | 453 | 450
years | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: AZ (Arimidex+Zoledronate) vs TZ (Tamoxifen+Zoledronate) vs AC (Arimidex Control) vs TC (Tamoxifen Control); To determine the effect of Zoledronic Acid (AZ and TZ) compared to no Zoledronic Acid (AC and TC) in terms of recurrence-free survival. Recurrence-free survival is defined as the time from randomization to the first occurrence of a local or regional recurrence, cancer in the contralateral breast, distant metastasis, second primary carcinoma, or death related to breast cancer; Test type: Superiority — No multiplicity adjustment was applied; p = 0.01, Log Rank; Cox Proportional Hazard = 0.65, 95% CI 2-sided [0.46 to 0.92]; From the Cox Proportional hazard model with Zoledronic Acid treatment fitted as a covariate. A hazard ratio < 1.0 indicates a lower average event rate and a longer recurrence-free time for Zoledronic Acid relative to no Zoledronic Acid

5. Secondary Outcome: Comparison of Anastrozole vs Tamoxifen in Premenopausal Patients With Non-metastatic Breast Cancer With Respect to Overall Survival (OS)
Description: OS is defined as time from randomization to death from any cause
Time Frame: as for outcome 1
Population: Intent-to-treat population: All participants assigned to one of the four treatment arms were included in the analysis
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
Number analyzed (Participants) | 450 | 450 | 453 | 450
years | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: AZ (Arimidex+Zoledronate) vs TZ (Tamoxifen+Zoledronate) vs AC (Arimidex Control) vs TC (Tamoxifen Control); To determine the effect of anastrozole (AZ and AC) compared to tamoxifen (TZ and TC) in terms of overall survival. Overall survival is defined as the time from randomization to death from any cause; Test type: Superiority — No multiplicity adjustment was applied; p = 0.07, Log Rank; Cox Proportional Hazard = 1.80, 95% CI 2-sided [0.96 to 3.38] — From the Cox Proportional hazard model with endocrine treatment fitted as a covariate. A hazard ratio > 1.0 indicates a higher average event rate and a shorter survival time for arimidex relative to tamoxifen

6. Secondary Outcome: Comparison of Zoledronate vs no Zoledronate in Premenopausal Patients With Non-metastatic Breast Cancer With Respect to Overall Survival (OS)
Description: OS is defined as time from randomization to death from any cause
Time Frame: as for outcome 1
Population: Intent-to-treat population: All participants assigned to one of the four treatment arms were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
Number analyzed (Participants) | 450 | 450 | 453 | 450
years | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events. | NA [NA to NA] — Not applicable, estimates cannot be calculated due to too few events.
Statistical Analysis 1: Comparison: AZ (Arimidex+Zoledronate) vs TZ (Tamoxifen+Zoledronate) vs AC (Arimidex Control) vs TC (Tamoxifen Control); To determine the effect of Zoledronic Acid (AZ and TZ) compared to no Zoledronic Acid (AC and TC) in terms of overall survival. Overall survival is defined as the time from randomization to death from any cause; Test type: Superiority — No multiplicity adjustment was applied; p = 0.10, Log Rank; Cox Proportional Hazard = 0.60, 95% CI 2-sided [0.32 to 1.11] — From the Cox Proportional hazard model with Zoledronic Acid treatment fitted as a covariate. A hazard ratio < 1.0 indicates a lower average event rate and a longer survival time for Zoledronic Acid relative to no Zoledronic Acid

ADVERSE EVENTS:
Time Frame: Maximum observation period per patient for all-cause mortality was 102 months starting with randomization. Reporting period for adverse events started with randomization and lasted until the first follow-up visit after the last treatment.
Description: All-cause mortality data presented for intention-to-treat analysis set and for the entire study. Serious adverse events (SAEs) reported during treatment phase plus 30 days, and after this period only if the investigator could not preclude a causal link to treatment with Anastrozole. Other adverse events were collected from randomization until the first follow-up visit after the last treatment.
Arm/Group | AZ (Arimidex+Zoledronate) | TZ (Tamoxifen+Zoledronate) | AC (Arimidex Control) | TC (Tamoxifen Control)
All-Cause Mortality (participants affected / at risk) | 9/450 | 7/450 | 18/453 | 8/450
Serious Adverse Events (participants affected / at risk) | 67/450 | 103/450 | 55/453 | 93/450
Other Adverse Events (participants affected / at risk) | 355/450 | 320/450 | 340/453 | 290/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZ (Arimidex+Zoledronate) (N=450) | TZ (Tamoxifen+Zoledronate) (N=450) | AC (Arimidex Control) (N=453) | TC (Tamoxifen Control) (N=450)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cutaneous reaction (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (6) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Disease of liver / gallbladder (Hepatobiliary disorders) | 2 (2) | 3 (4) | 2 (2) | 5 (6)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 7 (8) | 4 (4) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertonia (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Insult / TIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Irregular vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 5 (5) | 6 (6)
Lymphedema (arm, hand) (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Obstipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other tumors (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 2 (2) | 3 (3)
Ovarian changes (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve disease (Nervous system disorders) | 10 (13) | 1 (1) | 4 (5) | 4 (5)
Psychological disorder NOS (Psychiatric disorders) | 1 (1) | 3 (6) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 2 (2) | 2 (2) | 2 (3) | 0 (0)
Skin disease (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (9) | 3 (4) | 8 (8)
Spinal troubles/pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (5) | 5 (6) | 3 (5) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 5 (5) | 0 (0) | 3 (3)
Thyroid disease (Endocrine disorders) | 2 (3) | 0 (0) | 3 (3) | 3 (3)
Tinnitus/hearing loss (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Torn ligament/Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 3 (4)
Uro-genital tract infection (Infections and infestations) | 8 (9) | 7 (7) | 4 (4) | 6 (7)
Uterine polyp (Reproductive system and breast disorders) | 5 (6) | 52 (57) | 7 (7) | 39 (45)
Vaginal bleeding (Reproductive system and breast disorders) | 3 (3) | 13 (14) | 7 (7) | 6 (6)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZ (Arimidex+Zoledronate) (N=450) | TZ (Tamoxifen+Zoledronate) (N=450) | AC (Arimidex Control) (N=453) | TC (Tamoxifen Control) (N=450)
Arthralgia (Musculoskeletal and connective tissue disorders) | 150 (464) | 65 (133) | 112 (315) | 52 (124)
Bone pain (Musculoskeletal and connective tissue disorders) | 185 (571) | 132 (332) | 128 (439) | 94 (274)
Breast inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 9 (16) | 4 (6) | 3 (11) | 0 (0)
Cutaneous reaction (Skin and subcutaneous tissue disorders) | 15 (19) | 5 (7) | 18 (30) | 19 (28)
Diarrhea (Gastrointestinal disorders) | 12 (17) | 17 (21) | 11 (13) | 10 (13)
Dizziness (Nervous system disorders) | 18 (29) | 9 (14) | 7 (12) | 13 (19)
Fatigue (General disorders) | 98 (262) | 82 (179) | 93 (258) | 70 (156)
Fever (General disorders) | 46 (51) | 34 (38) | 11 (13) | 9 (11)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 9 (16) | 8 (12) | 6 (8) | 6 (11)
Headache (Nervous system disorders) | 85 (231) | 59 (117) | 63 (163) | 59 (155)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Hot flushes (Vascular disorders) | 25 (45) | 27 (50) | 25 (56) | 28 (43)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (10) | 0 (0) | 1 (3) | 0 (0)
Hypertonia (Nervous system disorders) | 25 (63) | 20 (36) | 20 (73) | 14 (29)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 3 (6) | 0 (0) | 0 (0)
Impaired vision (Eye disorders) | 29 (60) | 27 (58) | 22 (35) | 36 (84)
Incontinence (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Infection of ear, nose, or throat (Infections and infestations) | 5 (9) | 8 (15) | 5 (6) | 7 (12)
Irregular vaginal discharge (Reproductive system and breast disorders) | 2 (6) | 2 (2) | 2 (3) | 3 (10)
Leg edema (General disorders) | 2 (4) | 10 (15) | 2 (4) | 9 (17)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Lung inflammation (Respiratory, thoracic and mediastinal disorders) | 22 (32) | 9 (12) | 12 (14) | 13 (21)
Lymphedema (arm, hand) (Vascular disorders) | 26 (48) | 31 (63) | 28 (131) | 29 (64)
Morning stiffness (Musculoskeletal and connective tissue disorders) | 35 (72) | 14 (20) | 33 (90) | 11 (19)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (18) | 2 (2) | 9 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (17) | 6 (10) | 5 (6)
Nausea and vomiting (Gastrointestinal disorders) | 48 (88) | 29 (45) | 32 (56) | 23 (41)
Obstipation (Gastrointestinal disorders) | 0 (0) | 5 (11) | 1 (2) | 5 (7)
Other/minor (not categorized) (General disorders) | 119 (252) | 112 (219) | 107 (224) | 108 (212)
Ovarian changes (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Periodontal disease* (Gastrointestinal disorders) | 6 (11) | 3 (6) | 0 (0) | 5 (7)
Peripheral nerve disease (Nervous system disorders) | 29 (57) | 22 (36) | 14 (31) | 17 (30)
Psychological disorder NOS (Psychiatric disorders) | 80 (205) | 74 (197) | 97 (221) | 70 (174)
Sensory disturbance (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1) | 2 (4)
Skin disease (Skin and subcutaneous tissue disorders) | 26 (41) | 32 (68) | 16 (21) | 23 (32)
Spinal troubles/pain (Musculoskeletal and connective tissue disorders) | 16 (26) | 15 (30) | 15 (28) | 13 (26)
Stomach pain (Gastrointestinal disorders) | 17 (27) | 8 (13) | 13 (17) | 8 (12)
Tachycardia (Cardiac disorders) | 10 (16) | 9 (14) | 5 (7) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 (7) | 1 (2) | 4 (13) | 3 (5)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid disease (Endocrine disorders) | 5 (5) | 0 (0) | 2 (2) | 2 (2)
Tinnitus/hearing loss (Ear and labyrinth disorders) | 4 (5) | 1 (5) | 3 (3) | 2 (3)
Torn ligament/Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uro-genital tract infection (Infections and infestations) | 1 (1) | 7 (13) | 0 (0) | 3 (3)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 1 (1) | 5 (7)
Vaginal bleeding (Reproductive system and breast disorders) | 5 (6) | 4 (4) | 2 (3) | 5 (5)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 3 (12) | 2 (4) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 2 (5) | 2 (3) | 4 (10) | 2 (3)
Vaginal inflammation (Reproductive system and breast disorders) | 2 (4) | 4 (7) | 4 (5) | 8 (9)
Weight gain (Investigations) | 4 (7) | 7 (11) | 8 (12) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No